CLINICAL TRIAL: NCT06324383
Title: Enhancing Purpose and Well-Being Through a Volunteering Experience Connecting Veterans With English Language Learners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Piette, Professor of Health Behavior and Health Education, and of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1782599
Record Dates: First submitted 2024-03-12; First posted 2024-03-22 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety; Post Traumatic Stress Disorder
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Participants will be paired with an English language learner and engage in 8 weeks, 1 hour videoconferencing sessions.
  Interventions: Other: Intervention (videoconferencing)

INTERVENTIONS:
Other: Intervention (videoconferencing) — 1 hour videoconferencing sessions over 8 weeks with an English language learner partner.

SUMMARY:
The goal of this study is to refine and test a strategy for engaging Veterans with symptoms of depression, anxiety, and/or PTSD (Post Traumatic Stress Disorder) as volunteers to help English language learners (ELLs) improve their speaking skills via structured conversations using videoconferencing.

DETAILED DESCRIPTION:
The investigators goal is to do interventional research addressing the loss of purpose and social isolation among Veterans with depression and anxiety disorders. Following on the recent successful pilot among Veterans with depression, anxiety, and PTSD recruited via social media, the objective of this project is to conduct an intervention pilot with 40 pairs of Veterans with diagnosed depression, generalized anxiety disorder, and/or PTSD recruited from the VA, and English-language learners (ELLs). To accomplish this goal, staff will dedicate time in areas including: (1) Tailoring training and program materials for VA patients and English language learners (ELLs). (2) Enroll 40 pairs of Veterans and ELLs in the pilot. (3) Conduct orientation and supervised sessions via videocam for pilot participants. (4) Collect baseline/follow-up data including quantitative surveys and qualitative interviews of Veteran participants and ELLs. (5) Process and analyze pilot data. (6) Prepare an (Investigator Initiated Research) IIR as well as publication.

The intervention the investigators are developing is designed to have a national impact on the loss of purpose and social isolation among Veterans by evaluating a scalable, accessible, and safe strategy for increasing social engagement and volunteerism. The pilot the investigators propose will replicate a recent successful pilot conducted among Veterans with these conditions and recruited via social media (that project was approved by the University of Michigan's Health Sciences and Behavioral Sciences (HSBS) IRB (Institutional Review Board). The primary hypothesis is that structured contact between VA system users with mood and anxiety disorders and ELLs using accessible technology will enhance Veterans' sense of life purpose or "mattering" and improve mental health symptoms. The investigators hypothesize that satisfaction levels among Veterans recruited from VA and ELLs will be high, that the majority of both groups will have the intention of maintaining social contact after the study, and that ELLs will report improvements in their English-language confidence and fluency. The proposed intervention -V-SPEAK (Veterans Service Promoting English Acquisition and Knowledge), is highly scalable because it addresses the large unmet need for both Veteran volunteerism opportunities that are remote, removing barriers that traditional volunteer opportunities have; additionally, for individuals learning English as a second language, this program provides English practice among non-native English speakers in the US.

ELIGIBILITY:
Veteran coach participant

Inclusion Criteria:

* 18 years of age or older
* fluent English speakers
* diagnosis of depression, anxiety, or PTSD in their outpatient record in the last 12 months.
* be able to participate in a videoconference via a smartphone, tablet, laptop, or desktop computer in their home using a widely-accessible, no cost videoconferencing platform.

Exclusion Criteria:

* schizophrenia
* dementia
* traumatic brain injury that significantly impedes ability to participate in sessions
* significant sensory impairment
* current alcohol or drug abuse/dependence that would affect their ability to participate in the study

English Language Learner participant --

Inclusion Criteria:

* 18+ years of age
* be able to participate in a videoconference via a smartphone, tablet, laptop, or desktop computer in their home or referring organization using a widely-accessible, no cost videoconferencing platform
* basic ability to understand and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
France and Finney "Mattering" | Baseline, pre-intervention and Follow-up, immediately after 8-week intervention
  This is a 5 point scale where the minimum is 1 (strongly disagree) and maximum is 5 (strongly agree). Higher scores reflect higher mattering, and mattering is positively related to measures of well-being.
(Patient Health Questionnaire) PHQ-8 | Baseline, pre-intervention and Follow-up, immediately after 8-week intervention
  This is a 3 point scale (0= not at all, 3= nearly every day). Higher scores reflects greater depression.
(Generalized Anxiety Disorder) GAD-7 | Baseline, pre-intervention and Follow-up, immediately after 8-week intervention
  This is a 3 point scale (0= not at all, 3= nearly every day). Higher scores reflects greater anxiety.
(Posttraumatic Stress Disorder Checklist) PCL-5 | Baseline, pre-intervention and Follow-up, immediately after 8-week intervention
  PCL-5 is a 20-item self-report measure that assesses the 20 (Diagnostic and Statistical Manual) DSM-5 symptoms of PTSD. 5-point Likert (0 = "Not at all" to 4 = "Extremely"). Research on the PCL-5 suggested scores of 31 to 33 were optimally efficient for diagnosing PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — University of Michigan
Locations (1):
- Center for Clinical Management Research (CCMR), North Campus Research Complex, Ann Arbor, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT06324383/ICF_000.pdf